CLINICAL TRIAL: NCT00213395
Title: Clinical Efficacy of a Cephalic Mask for Noninvasive Ventilation During Acute Hypercapnic Respiratory Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004/015/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Acute Hypercapnic Respiratory Failure
Keywords: Noninvasive ventilation; Acute hypercapnic respiratory failure; Cephalic mask; Facial Mask
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

INTERVENTIONS:
Device: Interface for noninvasive ventilation

SUMMARY:
Noninvasive ventilation (NIV) is now a major therapeutic option to manage patients with acute hypercapnic respiratory failure (AHRF). Otherwise, patient-ventilator interfaces are determinant to get an optimal NIV efficacy in parallel with ventilatory comfort.

Facial masks during NIV are associated with deleterious consequences like gas leaks around the mask, skin breakdown (especially on the nasal bridge), claustrophobia and mask discomfort. In order to limit these side effects, a cephalic interface has been recently designed. Cephalic mask covers the whole anterior surface of the face and excessive mask fit pressure is therefore spread over a larger surface outside the nose area. However, this mask has a high volume that may interfere with NIV efficacy and may also induce claustrophobic sensations.

The aim of this study is to compare the clinical efficacy and tolerance of a cephalic mask versus a conventional oronasal mask during AHRF.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypercapnic respiratory failure
* Indication to noninvasive ventilation

Exclusion Criteria:

* Requirement for endotracheal intubation
* Proven pulmonary embolism
* Present or previous history of ophthalmologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Study Completion 2006-02

PRIMARY OUTCOMES:
Arterial blood gases

SECONDARY OUTCOMES:
Respiratory frequency
Severity scores
Ventilatory settings
Patient-ventilator adaptation
Tolerance
Outcome
Complications

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CUVELIER, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Pulmonary & Intensive Care Department - Rouen University Hospital,, Rouen, France